CLINICAL TRIAL: NCT01333813
Title: Long-term Antibody Persistence of Hepatitis B Antibodies and Immune Response to a Hepatitis B Vaccine (Engerix-B Kinder) Challenge in Children Previously Vaccinated With Infanrix Hexa Vaccine
Brief Title: Hepatitis B Antibody Persistence and Immune Response to Hepatitis B Vaccine Challenge in Previously Vaccinated Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112688
Record Dates: First submitted 2011-04-07; First posted 2011-04-12 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-08

CONDITIONS: Hepatitis B
Keywords: immune response; Engerix-B™Kinder; Persistence; challenge dose
MeSH Terms: conditions — Hepatitis B

ARMS (1):
- Engerix-B Kinder Group (Experimental): Subjects previously primed and boosted with 4 doses of Infanrix hexa vaccine in the first 2 years of life received a single dose of Engerix-B Kinder vaccine as an intramuscular (IM) injection into the deltoid region of the non-dominant arm at 7-8 years of age.
  Interventions: Biological: Engerix-B™ Kinder

INTERVENTIONS:
Biological: Engerix-B™ Kinder — Intramuscular, single dose

SUMMARY:
This study will evaluate the persistence of immunity to hepatitis B in healthy children aged 7 to 8 years, after previous vaccination with Infanrix hexa™ in the first two years of life, and also their ability to mount an immune response to the challenge dose of Engerix-B™ Kinder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* A male or female 7 to 8 years of age at the time of enrolment.
* Subjects with documented evidence of previous vaccination with four consecutive doses of Infanrix hexa™ as part of routine vaccination in Germany: three doses of primary vaccination received by 9 months of age and one booster dose received between 11 and 18 months of age.
* Written informed consent obtained from the parents/Legally Acceptable Representative(s) of the subject at the time of enrolment.
* In addition to the informed consent that will be signed by the parent(s)/Legally Acceptable Representative(s), written informed assent of the subject will be sought when the subject is judged able to understand by the investigator.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product, other than the study vaccine, within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous hepatitis B booster vaccination since administration of the fourth dose of Infanrix hexa™ booster in the second year of life.
* History of or intercurrent hepatitis B disease.
* Hepatitis B vaccination at birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before and ending 30 days after the hepatitis B vaccine challenge dose.
* Administration of immunoglobulins and/or any blood products within the three months preceding challenge dose or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the challenge dose of HBV vaccine.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the hepatitis B vaccine, or evidence of hypersensitivity after previous immunisation with a vaccine containing the hepatitis B component.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease and/or fever at the time of enrolment.

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2011-04-26; Primary Completion 2011-09-28 (Actual); Study Completion 2011-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Germany (12):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Kempten (Allgäu), Bavaria
  - GSK Investigational Site, Braunatal, Hesse
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112688 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112688 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112688 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112688 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112688 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112688 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 300 subjects were enrolled in the study. Among them 297 subjects were included in the Total Vaccinated cohort. Remaining 3 subjects were not included as they failed to meet protocol specified criteria and as such they are not included in the Participant Flow as Started.
Period: Overall Study
Arm/Group | Engerix-B Kinder Group
Started | 297
Completed | 297
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 297
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.5 (0.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144
  Male | 153

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-hepatitis B (Anti-HBs) Antibody Concentration Equal to or Above (≥) 100 Milli-International Units Per Milliliter (mIU/mL)
Description: A decrease in the specificity of the anti-HBs enzyme-linked immunosorbent assay (ELISA) had been observed in some studies for low levels of anti-HBs antibodies (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi-Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: One month (Month 1) after a challenge dose of Engerix-B Kinder vaccine
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects who had received a challenge dose of Engerix-B Kinder vaccine and for whom immunogenicity data were available at the post- Engerix-B Kinder challenge time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 262
Participants | 251

2. Secondary Outcome: Anti-HBs Antibody Concentrations After Previous Vaccination With Infanrix Hexa Vaccine.
Description: Antibody concentrations are expressed as Geometric mean antibody concentrations (GMCs) in mIU/mL.
  A decrease in the specificity of the anti-HBs ELISA had been observed in some studies for low levels of anti-HBs antibodies (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi-Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: Before (Day 0) a challenge dose of Engerix-B Kinder vaccine
Population: Analysis was performed on According-to-Protocol (ATP) cohort for persistence which included all subjects previously primed and boosted with 4 doses of Infanrix hexa in the first 2 years of life; with no evidence of hepatitis B infection or disease and for whom serological results were available at the pre- Engerix-B Kinder challenge time point.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 287
mIU/mL | 36.6 [29.7 to 45.1]

3. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations Equal to or Above the Protocol Specified Cut-off Values After Previous Vaccination With Infanrix Hexa Vaccine
Description: Anti-HBs antibody concentrations cut-off values assessed were ≥ 6.2 mIU/mL (previously 3.3 mIU/mL), ≥ 10 mIU/mL, ≥ 10 mIU/mL to <100 mIU/mL and ≥ 100 mIU/mL. A decrease in the specificity of the anti-HBs ELISA had been observed in some studies for low levels of anti-HBs antibodies (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi-Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis and the initial 3.3 mIU/mL seropositivity cut-off was revised into the new 6.2 mIU/mL cut-off.
Time Frame: Before (Day 0) a challenge dose of Engerix-B Kinder vaccine
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 287
Participants
  Anti-HBs antibody ≥ 6.2 mIU/mL | 225
  Anti-HBs antibody ≥ 10 mIU/mL | 207
  Anti-HBs antibody between ≥ 10 and < 100 mIU/mL | 118
  Anti-HBs antibody ≥ 100 mIU/mL | 89

4. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations Equal to or Above Protocol Specified Cut-off Values
Description: Anti-HBs antibody concentrations cut-off values assessed were ≥ 6.2 mIU/mL (previously 3.3 mIU/mL) and ≥ 10 mIU/mL. A decrease in the specificity of the anti-HBs ELISA had been observed in some studies for low levels of anti-HBs antibodies (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi-Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis and the initial 3.3 mIU/mL seropositivity cut-off was revised into the new 6.2 mIU/mL cut-off.
Time Frame: One month (Month 1) after a challenge dose of Engerix-B Kinder vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 262
Participants
  Anti-HBs antibody ≥ 6.2 mIU/mL | 259
  Anti-HBs antibody ≥ 10 mIU/mL | 259

5. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations are expressed as Geometric mean antibody concentrations (GMCs) in mIU/mL. A decrease in the specificity of the anti-HBs had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi-Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: One month (Month 1) after a challenge dose of Engerix-B Kinder vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 282
mIU/mL | 4819.1 [3749.7 to 6193.6]

6. Secondary Outcome: Number of Subjects Demonstrating an Anamnestic Response to the Engerix-B Kinder Challenge Dose
Description: The anamnestic response is defined as an antibody concentration ≥ 10 mIU/mL at post Engerix-B Kinder challenge dose time point for initially seronegative subjects ,and as an antibody concentration at post Engerix-B Kinder challenge dose time point ≥ 4 fold the pre-vaccination antibody concentration for initially seropositive subjects. A seropositive/seronegative subject was defined as subject with HBs antibody concentration below/greater than or equal to the seropositivity cut-off of 6.2 mIU/mL. A decrease in the specificity of the anti-HBs ELISA had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis and the initial 3.3 mIU/mL seropositivity cut-off was revised into the new 6.2 mIU/mL cut-off.
Time Frame: After Engerix-B Kinder challenge dose (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 262
Participants | 253

7. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was occurrence of any local symptom regardless of their intensity grade. Grade 3 pain was considerable pain at rest that prevented normal everyday activities. Grade 3 redness and swelling was > 50 millimeter (mm).
Time Frame: During the 4-day (Day 0-3) follow-up period after the challenge dose of Engerix-B Kinder vaccine
Population: Analysis was performed on Total Vaccinated cohort which included all subjects who received the challenge dose of Engerix-B Kinder vaccine .
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 297
Participants
  Any pain | 91
  Grade 3 pain | 2
  Any redness | 84
  Grade 3 redness | 0
  Any swelling | 49
  Grade 3 swelling | 0

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache and temeperature.
  Any temperature was defined as axillary temperature ≥ 37.5 degree centigrade (°C), grade 3 temperature was axillary temperature > 39.0°C. For other symptoms, any was defined as occurrence of any general symptom regardless of intensity grade or relation to vaccination and grade 3 was defined as a general symptom that prevented normal activity. Related was a general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period after the challenge dose of Engerix-B Kinder vaccine
Population: Analysis was performed on Total Vaccinated cohort which included all subjects who received the challenge dose of Engerix-B Kinder vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 297
Participants
  Any fatigue | 37
  Grade 3 fatigue | 1
  Related fatigue | 21
  Any gastrointestinal symptoms | 27
  Grade 3 gastrointestinal symptoms | 5
  Related gastrointestinal symptoms | 5
  Any headache | 36
  Grade 3 headache | 2
  Related headache | 15
  Any temperature | 14
  Grade 3 temperature | 0
  Related temperature | 11

9. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-30) follow-up period after the challenge dose of Engerix-B Kinder vaccine
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 297
Participants | 42

10. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination.
Time Frame: After the challenge dose of Engerix-B Kinder vaccine up to the study end (Day 0 to Month 1)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 297
Participants | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from Day 0 to Month 1. Systematically assessed frequent adverse events were assessed during the 4-day post vaccination period.
Arm/Group | Engerix-B Kinder Group
Serious Adverse Events (participants affected / at risk) | 2/297
Other Adverse Events (participants affected / at risk) | 164/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B Kinder Group (N=297)
Hypersensitivity (Immune system disorders) | 1
Lyme disease (Infections and infestations) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B Kinder Group (N=297)
Pain (General disorders) | 91
Redness (General disorders) | 84
Swelling (General disorders) | 49
Fatigue (General disorders) | 37
Gastrointestinal symptoms (General disorders) | 27
Headache (General disorders) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.